CLINICAL TRIAL: NCT06584591
Title: Neuromodulation-Enhanced Use of RObotic Balance Training to Improve Postural Control in Individuals With Traumatic Brain Injury
Brief Title: NEUROBALANCE Training to Improve Postural Control in Individuals With Traumatic Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vikram Shenoy Handiru, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-1261-24
Record Dates: First submitted 2024-09-02; First posted 2024-09-05 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Brain Injury; TBI; Diffuse Axonal Brain Injury; Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries, Diffuse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The mode of HD-tDCS (active/sham) will be masked for the participant and outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- RBT + Active HD-tDCS Group (Experimental): Participants will engage in balance and postural control training on a robotic balance platform called Hunova (Movendo, Italy). Before balance training, the current intensity of 2 mA will be delivered to the leg motor area identified using neuronavigated transcranial magnetic stimulation, and the stimulation will be turned ON for 20 minutes.
  Interventions: Device: Combined (Robotic balance training and high-definition transcranial direct current stimulation)
- RBT + Sham HD-tDCS Group (Sham Comparator): Participants will engage in balance and postural control training on a robotic balance platform called Hunova (Movendo, Italy). Before balance training, the current intensity of 2 mA will be delivered to the leg motor area identified using neuronavigated transcranial magnetic stimulation, and the stimulation will be turned ON transiently for 30 s, to provide a sensation of stimulation.
  Interventions: Device: Combined (Robotic balance training and high-definition transcranial direct current stimulation)
- SOC Control Group (Other): The SOC control group participants will perform conventional physical therapy exercises delivered by a trained PT.
  Interventions: Other: Standard of Care Balance Training

INTERVENTIONS:
Device: Combined (Robotic balance training and high-definition transcranial direct current stimulation) — The robotic platform will train the participants to maintain dynamic balance in the sagittal and the transverse planes (mediolateral and anterior-posterior directions) and engage in core stability and trunk control with seated balance exercises. In addition, high-definition transcranial direct current stimulation (HD-tDCS) will be used as an adjuvant to robotic balance training by priming the corticospinal circuits.
  Arms: RBT + Active HD-tDCS Group; RBT + Sham HD-tDCS Group
Other: Standard of Care Balance Training — Participants in this group will receive a standard-of-care balance training administered by the Physical therapist.
  Arms: SOC Control Group

SUMMARY:
Our proposed study, "NEUROBALANCE," aims to evaluate the effectiveness of a combined intervention involving robotic balance training and noninvasive brain stimulation in improving balance functions in individuals with chronic traumatic brain injury (TBI). The study will recruit 45 participants who have had a TBI for over six months and experience persistent balance deficits. Participants will be randomized into three groups: (1) robotic balance training with active brain stimulation, (2) robotic balance training with sham brain stimulation, and (3) standard-of-care rehabilitation.

The study will involve 12 training sessions over four weeks, with assessments conducted at baseline, post-training, and two months post-training to evaluate balance recovery and retention. The primary focus is understanding how this intervention affects brain and muscle activity during balance tasks and how these changes translate into functional improvements in clinical outcome measures of balance function. Additionally, participant feedback on brain stimulation and exercise engagement will be collected to inform future studies.

This research is particularly relevant to military service members, as TBI and balance impairments are common among this population. The findings may guide the development of personalized training protocols and contribute to broader rehabilitation strategies.

DETAILED DESCRIPTION:
Background: Traumatic Brain Injury (TBI) is one of the severe health conditions with debilitating consequences, affecting more than 2.5 million individuals in the US alone. Balance dysfunction is one of the most disabling outcomes of TBI, affecting roughly half of those who have TBI even after ten years have passed after their accident, and further, it increases the risk of falls due to poor postural control. The current challenges are that there are currently no well-established rehabilitation treatments that have been shown to have long-term retention of balance recovery in TBI survivors with chronic balance complaints. Therefore, we need novel therapeutic strategies using rehabilitation engineering that can target sensorimotor integration and improved proprioceptive control to improve balance function, thereby alleviating the long-term burden on TBI survivors and their caregivers.

Hypothesis and Rationale: We hypothesize that the balance and postural control recovery requires a multimodal strategy, and we propose robotic balance training (RBT) using the Hunova platform (Movendo Technology, Italy), as it has an advantage of supporting dynamic balance in not only sagittal plane but also transverse plane (mediolateral and anterior-posterior directions), and allows for core stability and trunk control with its unique seated balance exercises. In addition, we hypothesize that by using high-definition transcranial direct current stimulation (HD-tDCS) as an adjuvant to RBT, HD-tDCS will facilitate top-down neuromuscular control of balance through corticospinal circuits, whereas the robotic platform will enable bottom-up feedback of response to platform perturbations. Overall, we anticipate that the combined intervention will improve reactive and anticipatory postural control, position sense, and proprioceptive control, gain lower-limb strength, increase ankle range of motion, and stimulate attention through game-like exercises.

Study Design: We propose a single-center, investigator-blinded, randomized, sham-controlled triple-arm parallel-group, superiority trial study. Forty-five adult individuals with chronic TBI with complaints of balance dysfunction (injury onset > 6 months before screening) will be randomized into one of the three groups: (1) Real HD-tDCS + RBT, (2) Sham HD-tDCS + RBT, and (3) Control group receiving dose-matched standard of care rehabilitation treatment. All participants will undergo 12 sessions (3 days × 4 weeks) of intervention. A total of 3 assessment visits (before training, immediately after 4-week training, and 2-months after the last training visit) will be conducted to evaluate the functional recovery and neurophysiological changes due to intervention.

Specific Aim-1: To determine whether there is an overall treatment effect of targeted neuromodulation combined with robotic balance training on balance outcomes immediately after 4-week training function in people with TBI. The change in Berg Balance Scale score from baseline to 4-week post-training will be the primary outcome measure. The secondary outcome measures of balance recovery will be the changes in Mini BESTest, Functional Gait Assessment, and Trunk Impairment Scale scores from baseline to 4-week post-training. We hypothesize that the Real HD-tDCS + RBT will show the largest improvement in the balance outcomes.

Secondary Aim-2: To characterize the top-down and bottom-up neurophysiological mechanisms of balance control due to neuromodulation-enhanced robotic training. We will measure the neurophysiological outcomes of EEG and EMG activity, and posturography outcomes of body sway during platform perturbation task at baseline, 4-week post-training, and 2-month follow-up. Specifically, the intervention-induced changes in the cortical reactivity amplitude, muscle coactivation, and center of displacement will be compared across groups.

Secondary Aim-3: To study the association between the intervention-related changes in the balance function endpoints and graph-theoretic measures of cortical functional connectivity. We will use a multivariate statistical approach-partial least squares correlation-to identify a latent component that characterizes the correlation between the 4-week intervention-related changes in balance outcome measures and EEG corticocortical functional connectivity features measured during platform perturbation task.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18-75 years
2. Diagnosed with a non-penetrating TBI at least six months before the screening.
3. Have complaints of impaired balance and poor postural control determined by a BBS score of ≤50.
4. Ability to stand upright with or without support for at least 20 seconds
5. Ability to walk with or without a walking aid for at least ten meters
6. Not planning to change medication in the next four months
7. Minimum Cognitive Ability to understand the verbal instructions and comply with the study procedures, as determined by the University of California, San Diego, Brief Assessment of Capacity to Consent Instrument (UBACC).

Exclusion Criteria:

1. Currently undergoing any regular physical therapy program or research studies focusing on balance functions.
2. Having a stroke or a penetrating TBI.
3. Affected by the peripheral nerve injury, neuromuscular conditions, or orthopedic issues of lower limbs before TBI, or have any persistent pain or difficulty maintaining blood pressure while upright.
4. Have a scalp or skin condition (e.g., psoriasis or eczema) on the scalp near the stimulation site.
5. Severe visual impairment (e.g., spatial neglect) or hearing problems may affect study compliance.
6. Any other neurological injury or psychiatric conditions (e.g., severe anxiety or schizophrenia, etc.)
7. Not being pregnant or thinking of becoming pregnant during the study period.
8. Diagnosed with alcohol or substance abuse in the last three years.
9. Contraindications to TMS, including the presence of metallic implants in the head and history of seizures or medication-resistant epilepsy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | Baseline, post 4-week training, 2-month follow-up
  A widely used outcome measure of static standing balance function (Newstead et al., 2005), categorized under the 'Activity' subsection of ICF domain. BBS scores range from 0 to 56 (the higher, the better). The change in BBS scores from baseline to 4 weeks post-training will be the primary endpoint.

SECONDARY OUTCOMES:
Functional Gait Assessment (FGA) | Baseline, post 4-week training, and 2-month follow-up
  To assess dynamic balance during walking, unlike BBS, it is not prone to the ceiling effect(Van Bloemendaal et al., 2019). FGA will be used as the secondary outcome measure of balance function and gait. FGA comes under the ICF domains of 'Activity' and 'Body Function.'
Mini Balance Evaluation Systems Test (MBT) | Baseline, post 4-week training, and 2-month follow-up
  To identify the risk of falls (Yingyongyudha et al., 2016) with a high internal consistency with BBS and similar advantage of FGA, i.e., no ceiling effect. MBT will be used as the secondary endpoint of the balance function.
Trunk Impairment Scale (TIS) | Baseline, post 4-week training, and 2-month follow-up
  To estimate the trunk motor impairment(Verheyden et al., 2004). The scale ranges from 0 to 23 and assesses static and dynamic postural control.
Center of Pressure (COP) Displacement | Baseline, post 4-week training, and 2-month follow-up
  To evaluate the body sway in response to the perturbations of the posturography platform.
TMS-evoked EEG Potentials (TEP) | Baseline, post 4-week training, and 2-month follow-up
  A neurophysiological outcome measure of cortical reactivity. TEPs can directly measure cortical reactivity without being affected by the distal components of the nervous system, especially in neurological populations(Keser et al., 2022). In contrast to motor-evoked potentials, TEPs also offer the advantage of eliciting cortical responses at TMS intensity below the resting motor threshold.
EEG Corticocortical Functional Connectivity | Baseline, post 4-week training, and 2-month follow-up
  The imaginary part of coherence (iCOH) measured from the source-space EEG time-series will be used as an outcome measure of corticocortical connectivity, representing sensorimotor functional integration.
EEG-to-EMG Corticomuscular Connectivity | Baseline, post 4-week training, and 2-month follow-up.
  EEG-to-EMG directed transfer function (DTF) will be used as an outcome measure of causal information flow from cortical areas to the leg muscles (Artoni et al., 2017; Peterson & Ferris, 2019). This measure is intended to capture changes in the efferent communication due to combined interventions.
EMG Muscle Coactivation | Baseline, post 4-week training, and 2-month follow-up.
  EMG co-contraction index will be used as an outcome measure of muscle activation between the antagonist and agonist muscle pair involved in reactive balance control.
Quality of Life after Brain Injury (QOLIBRI) | Baseline, post 4-week training, and 2-month follow-up.
  A 37-item questionnaire to assess the level of satisfaction with different aspects of Quality of Life (QoL), on a scale of 1 (not at all satisfied) to 5(very satisfied); QOLIBRI is categorized under the ICF domain of 'Participation.'
Physical Activity Enjoyment Scale (PACES) | Post 4-week training
  An 18-item questionnaire with a 7-point Likert scale (higher scores represent increased activity enjoyment) has high reliability and validity(Murrock et al., 2016). The PACES scores will be used during training to assess the enjoyability of the balance exercises.
Dizziness Handicap Inventory (DHI) | Baseline, post 4-week training, and 2-month follow-up.
  A 25-item questionnaire with a 3-point scale to evaluate how dizziness or unsteadiness has affected daily activities in the last month. (Jacobson & Newman, 1990).

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Shenoy Handiru, Ph.D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
We will submit the IPD available in the tabular data to the Open Data Commons for Traumatic Brain Injury (ODC-TBI) after removing any personal or private identifiers. The neurophysiological data (such as the EEG, TMS, and EMG) will be shared on OpenNeuro.org (or a similar platform) in a BIDS-standardized format.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Six months after study completion.
Access Criteria: "Authorized Users" (i.e., all Users with an account on the ODC-TBI) will have access to the data.
URL: http://odc-tbi.org